CLINICAL TRIAL: NCT02936908
Title: Modalities of Respiratory Care, Vital and Respiratory Prognosis in Neuromuscular Patients Admitted to an Intensive Care Unit for Respiratory Failure
Brief Title: Respiratory Care in Intensive Care Unit for Neuromuscular Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0558
Record Dates: First submitted 2016-08-19; First posted 2016-10-18 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Respiratory Failure
Keywords: Neuromuscular Diseases; Muscular dystrophy; Amyotrophic Lateral Sclerosis; Acute respiratory failure; respiratory care; mechanical ventilation; weaning; Intensive Care Unit; Critical Care; Survival
MeSH Terms: conditions — Respiratory Insufficiency; Neuromuscular Diseases; Muscular Dystrophies; Amyotrophic Lateral Sclerosis | interventions — Interactive Ventilatory Support

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ventilatory support: Adult patients presenting a neuromuscular disease, with involvement of respiratory or bulbar muscles
  Interventions: Other: Ventilatory support

INTERVENTIONS:
Other: Ventilatory support — Initiation of mechanical ventilatory support, invasive or non-invasive, Or modification of mechanical ventilatory support (modification of the parameters of the device, change of material, switch from non-invasive to invasive)

SUMMARY:
Retrospective multicentric observational study exploring the population of adult neuromuscular patients presenting a respiratory distress requiring their admission in an Intensive Care Unit (ICU) for ventilatory support.

Research of markers associated with long term mortality and ventilatory status.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years old
* First stay in a ICU ward
* Inclusion period : Admission in ICU between 01/01/2007 and 31/12/2015
* Presenting an acute respiratory distress at admission or during ICU stay
* Diagnosis of neuromuscular disease confirmed before Hospital discharge

Exclusion Criteria:

* Absence of respiratory failure during ICU stay (ICU stay for monitoring or for a specialized invasive procedure in the absence of respiratory failure, for example)
* Neuromuscular disease not proven or uncertain diagnosis
* Anterior admission in ICU ward for vital organ failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting a neuromuscular disease, with involvement of respiratory or bulbar muscles.
  Neuromuscular diseases concerned :
  Central or Peripheral metabolic, toxic, or inflammatory neuropathies, Central or peripheral neurodegenerative or hereditary disorders Myopathies, amongst them dystrophinopathies, myotonic dystrophies Myasthenia gravis Tetraplegy, consequence of cervical spinal cord injury
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Mortality | until 2016.12.31
  number of death

SECONDARY OUTCOMES:
Definitive long term invasive ventilatory support | until 2016.12.31
  Date of tracheotomy for definitive long term invasive ventilatory support
Mortality attributable to a respiratory issue | until 2016.12.31
  For patients for which this information is available, cause of death described as reliable to a respiratory issue in any medical document available.
Re-hospitalization in a ICU-Ward | until 2016.12.31
  clinical deterioration requiring a new hospitalization in a ICU ward, after first hospitalization discharge.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHU Clermont Ferrand, Clermont-Ferrand
  - CHU Grenoble, Grenoble
  - Hôpital de la Croix Rousse, Lyon
  - Hôpital Nord CHU St Etienne, Saint-Etienne